CLINICAL TRIAL: NCT03439215
Title: PF-06463922 for Crizotinib Pretreated ROS1 Positive Non-small-cell Lung Cancer: a Phase II Trial (PFROST)
Brief Title: PF-06463922 for Crizotinib Pretreated ROS1 Positive Non-small-cell Lung Cancer
Acronym: PFROST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione Ricerca Traslazionale (Other)
Collaborators: Clinical research technology Srl (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FoRT 01/2016
Record Dates: First submitted 2018-02-01; First posted 2018-02-20 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: ROS1 positive; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lorlatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lorlatinb Arm (Experimental): Eligible patients will be treated with Lorlatinib at the dose of 100 mg QD p.o.
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — Lorlatinib is a novel small-molecule ROS1/ALK inhibitor that was optimized for robust brain penetration.
  Other Names: Lorlatinb

SUMMARY:
This is a phase II study assessing response rate to PF-06463922 in patients with ROS1 translocation resistant to previous crizotinib therapy. Eligible patients will be treated with the study drug until disease progression, unacceptable toxicity or patient refusal. Disease assessment will be performed every 8 weeks according to RECIST criteria.

DETAILED DESCRIPTION:
PF-06463922 is a novel small-molecule ROS1/ALK inhibitor that was optimized for robust brain penetration. The results showed that PF-06463922 is most potent against ROS1 and ALK, with selectivity ratios >100-fold for ROS1 over the 204 kinases tested. A recent study has investigated the activity of PF-06463922 against the crizotinib-resistant ROS1G2032R mutation in both recombinant enzyme and cell-based assays. PF-06463922 effectively inhibited the catalytic activity of recombinant ROS1G2032R and the CD74-ROS1G2032R fusion kinase in BaF3 cells. This effect translated directly into an antiproliferative response. These results, together with its exquisite ROS1 potency and ability to suppress the resistant ROS1 mutations, supports the clinical evaluation of PF-06463922 in ROS1-positive NSCLC, including patients who have developed resistance to crizotinib because of the acquired G2032R mutation and/or brain metastases.

This is a phase II study assessing response rate to PF-06463922 in patients with ROS1 translocation resistant to previous crizotinib therapy. Eligible patients will be treated with the study drug until disease progression, unacceptable toxicity or patient refusal. Disease assessment will be performed every 8 weeks according to RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent;
2. Male or female patient ages ≥ 18 years;
3. Histologically/cytologically confirmed diagnosis of NSCLC with evidence of ROS1 rearrangement;
4. Possibility to perform a new tumor biopsy or tumor tissue collected at the time or after crizotinib failure;
5. Patient pretreated with crizotinib with evidence of disease progression during crizotinib therapy;
6. At least one radiological measurable disease according to RECIST criteria;
7. At least 1 previous standard chemotherapy regimen;
8. Performance status 0-2 (ECOG);
9. Patient compliance to trial procedures
10. Adequate bone marrow function (ANC ≥ 1.5x109/L, platelets ≥ 100x109/L, haemoglobin > 9 g/dl);
11. Adequate liver function (bilirubin < grade 2, transaminases no more than 3xULN/<5xULN in present of liver metastases);
12. Normal level of alkaline phosphatase and creatinine;
13. If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of approved contraceptive method [intrauterine contraceptive device (IUD), birth control pills, or barrier device] during and for ninety (90) days after end of treatment.

Exclusion Criteria:

1. No ROS1 rearrangement 2. No previous therapy with crizotinib; 3. No evidence of crizotinib failure; 4. No post-crizotinib tumor tissue available; 5. Absence of any measurable lesions; 6. No previous chemotherapy; 7. Concomitant radiotherapy or chemotherapy; 8. Symptomatic brain metastases; 9. Diagnosis of any other malignancy during the last 5 years, except for in situ carcinoma of cervix uteri and squamous cell carcinoma of the skin; 10. Predisposing factors for acute pancreatitis (e.g., uncontrolled hyperglycaemia, current gallstone disease, alcoholism); 11. History of extensive disseminated/bilateral or known presence of Grade 3 or 4 interstitial fibrosis or interstitial lung disease including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis and pulmonary fibrosis (but not history of prior radiation pneumonitis); 12. Pregnancy or lactating female; 13. Other serious illness or medical condition potentially interfering with the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-13 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Response rate to PF-06463922 in patients with ROS1 translocation resistant to crizotinib | From date of the first enrolment until the date of last documented progression or date of death from any cause, assessed up to 36 months
  Response rate to PF-06463922 in patients with ROS1 translocation resistant to crizotinib

SECONDARY OUTCOMES:
Progression-free survival (PFS), The length of time during and after the treatment of a disease,that a patient lives with the disease but it doesn't get worse. | From date of the first enrolment until the date of last documented progression or date of death from any cause, assessed up to 36 months
  Progression-free survival (PFS) will be calculated from the time between the baseline/start of treatment visit to the time of first occurrence of progressive disease (PD) or death from any cause. Patients who have neither progressed nor died at time of analysis will be censored at the date of last tumor assessment where non progression was documented (i.e. CR, PR or SD)
Overall Survival (OS): Time from the start of treatment until death from any cause | From date of the first enrolment until the date of last documented progression or date of death from any cause, assessed up to 36 months
  Overall survival (OS) will be calculated from the time between the baseline/start of treatment visit to the date of death, irrespective of the cause of death. Patients still alive at the time of analysis will be censored at the date they were last known to be alive
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From date of the first enrolment until the date of last documented progression or date of death from any cause, assessed up to 36 months
  Patients will be closely monitored for signs and symptoms of potential adverse events, and will undergo frequent laboratory tests to assess lipids, pancreas, liver, kidney, and haematological function.
Correlation with additional tumor biomarkers in tumor tissue or blood | From date of the first enrolment until the date of last documented progression or date of death from any cause, assessed up to 36 months
  Correlation with additional tumor biomarkers in tumor tissue or blood

CONTACTS AND LOCATIONS:
Locations (20):
- Italy (20):
  - IRCCS - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST)- Oncologia Medica, Meldola, Forlì- Cesena
  - Sacro Cuore- Don Calabria Hospital- U.O.C. Oncologia Medica, Negrar, Verona
  - Istituto Toscano Tumori Ospedale San Donato- U.O.C. di Oncologia Medica Dipartimento di Oncologia USL-8, Arezzo
  - Azienda Ospedaliera di Rilievo Nazionale "S.G. Moscati", Avellino
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - IRCCS A.O.U. San Martino- IST- Istituto Nazionale per la Ricerca sul Cancro- U.O.S. Tumori Polmonari, Genova
  - Istituto Europeo di Oncologia - Divisione di Oncologia Toracica, Milan
  - A.O.U. Policlinico di Modena- Oncologia Ematologia e Malattie Apparato Respiratorio, Modena
  - A.O. San Gerardo, Monza
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Istituto Oncologico Veneto IRCCS- UOS Oncologia Toracica UOC. Oncologia Medica 2, Padua
  - Casa di Cura La Maddalena- U.O. Oncologia medica, Palermo
  - Azienda Ospedaliera Universitaria di Parma- Struttura Complessa di Oncologia Medica, Parma
  - Azienda Ospedaliera di Perugia- S.C. Oncologia Medica, Perugia
  - Ospedale di Ravenna- Oncologia Medica, Ravenna
  - Ospedale "Infermi" Rimini, Rimini
  - ASST della Valle Olona - Ospedale di Saronno, Saronno
  - A.O.U. San Luigi Gonzaga, Torino
  - Azienda ULSS 9 TREVISO-UOC Oncologia Medica, Treviso
  - Policlinico 'G.B.Rossi' Borgo Roma - A.O.U. Integrata (Giampaolo Tortora)- Oncologia Medica, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PFROST trial — https://www.cr-technology.com/fort/?studio_clinico=pfrost